CLINICAL TRIAL: NCT06174207
Title: Hyperoxia During Pulmonary Rehabilitation in Chronic Lung Disease - Does it Matter?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Switzerland University of Applied Sciences (Other)
Collaborators: University Hospital, Zürich (Other); Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RehaExO2
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma; Pulmonary Hypertension; Interstitial Lung Disease; Chronic Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Hypertension, Pulmonary; Lung Diseases, Interstitial | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Start with Constant Work Rate Exercise Test with 5l/min room air applied via nasal cannula.
  Interventions: Other: Oxygen
- Experimental Group (Experimental): Start with Constant Work Rate Exercise Test with 5l/min Oxygen Therapy applied via nasal cannula.
  Interventions: Other: Oxygen

INTERVENTIONS:
Other: Oxygen — Standard supplemental Oxygen therapy (5l/min) will be applied with an oxygen concentrator via nasal cannula.

SUMMARY:
Chronic respiratory diseases are a global burden. Treatment options have improved in recent years, pulmonary rehabilitation plays a key role. Oxygen therapy is recommended in patients with a low saturation at rest, but no clear guidance is given for patients who desaturate during exercise. The effect of ambulatory oxygen during exercise is not yet completely understood, especially in those patients with exercise-induced desaturation.

Aim: The goal of this study is to analyse the effect of supplemental oxygen given during a constant work rate exercise test (CWRET) on a cycle ergometer compared to sham air.

Methods: We plan to include 25 Patients respiratory patients undergoing pulmonary rehabilitation (male and female; aged >18 years; stable condition >3 weeks (e.g. no exacerbations); resting oxygen saturation (SpO2) ≥ 88%) with exercise induced hypoxemia defined by a fall in oxygen saturation by ≥ 4% during a 6-minute walking test. Patients will undergo an incremental exercise test with a ramp protocol (for evaluating the maximal workload) and two CWRET (75% of the maximal workload) with ambulatory oxygen or placebo (sham air) via standard nasal canula at a flow rate of 5l/min. Patients and assessors will be blinded. The difference endurance time of the CWRET with oxygen vs. sham air will be the primary outcome of this study.

Data will be summarized by means (SD) and medians (quartiles) for normal and non-normal distributions. Effects of treatment will be evaluated by mean differences with 95% confidence intervals, T-tests or Wilcoxon matched pair tests as appropriate. A p-value threshold of <0.05 or a confidence interval not including zero will be considered as statistically significant. Analyses will be performed according to the intention to treat principle.

ELIGIBILITY:
Inclusion Criteria:

* We will include male and female lung disease patients undergoing pulmonary rehabilitation: aged ≥ 18 years; stable condition > 3 weeks (e.g. no exacerbations); resting oxygen saturation (SpO2) ≥ 88% and exercise induced hypoxemia defined by a fall in SpO2 by ≥ 4% during a 6-minute walking test (6MWT); informed consent as documented by signature.

Exclusion Criteria:

* Severe daytime resting hypoxemia (SpO2 < 88% or partial pressure of oxygen (PaO2) < 8 kPa); unstable condition requiring adaptation of pharmacologic and other treatment modalities or requirement of intensive care or relevant severe concomitant disease; inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, neurological or orthopedic problems with walking disability or inability to ride a bicycle; women who are pregnant or breast feeding; enrolment in another clinical trial with active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Constant Work Rate Exercise Test | 7 days
  Endurance time measured with Constant Work Rate Exercise Test (CWRET) (75% of the maximal work rate from the maximal ramp exercise test)

SECONDARY OUTCOMES:
SpO2 | 7 days
  SpO2 by finger pulse oximetry, brain and muscle tissue oxygenation by near infrared spectroscopy (NIRS) at rest and end-exercise CWRET
Heart Rate | 7 days
  Heart rate at rest and end-exercise CWRET
Borg Scale (0-10) | 7 days
  Borg scale (dyspnoea and fatigue) at rest and end-exercise CWRET
Blood Pressure | 7 days
  Blood pressure at rest and end-exercise CWRET

CONTACTS AND LOCATIONS:
Overall Officials: Swantje Beyer, Dr.med., Principal Investigator — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No